CLINICAL TRIAL: NCT01336309
Title: Development of a Translational Tool to Study Yoga Therapy
Status: Completed | Type: Observational
Sponsor: University of Connecticut (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Crystal Park, Professor, University of Connecticut
Other Study IDs: IRB # H10-226; 1R01AT006466-01 (NIH)
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Health Behavior
Keywords: Yoga
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Focus Group: We conducted three focus groups per site, at three sites, with around eight people each. These data were used to guide refinement and selection of the items we developed for Phase III data collection. We will administer the Yoga Research Tool.
  Interventions: Behavioral: Yoga Research Tool
- Cognitive Interviews: We conducted cognitive interviews at three different sites, with about ten in each group. These data were used to guide refinement and selection of the items we developed for Phase III data collection. We collected this data via a large, online survey and administered the Yoga Research Tool.
  Interventions: Behavioral: Yoga Research Tool
- Survey Prototype Administration: We administered a prototype of the study measure to a large group of yoga students, with about 450 total participants. These data were used to further inform the refinement and selection of items to be used in the final measure.
  Interventions: Behavioral: Yoga Research Tool
- Reliability and Validity Testing: We are conducting yoga classes at community partner facilities near each site, with about ten participants in each class. Participants at each class will complete the study measure and related questionnaires, in order to test the reliability and validity of the study measure.
  Interventions: Behavioral: Yoga Research Tool

INTERVENTIONS:
Behavioral: Yoga Research Tool — We will be collecting data from a literature search, focus groups, cognitive interviews, and an online survey to build a measure for yoga researchers.

SUMMARY:
This study comprises 4 phases designed to systematically develop and test a reliable, valid and useful quantitative measure of the components and dimensions of yoga; each phase builds on the previous phase. Phase I aims to gain a comprehensive understanding of the relevant aspects of yoga therapy and develop a large pool of potential questionnaire items by conducting a thorough literature review and focus groups with yoga teachers and students. These data will be analyzed using rigorous qualitative methods to identify key conceptual dimensions associated with yoga interventions. Phase II will develop a prototypic questionnaire to assess yoga therapy by refining and honing information from Phase I and conducting cognitive interviews to further develop this instrument. Phase III will pilot test the measure in a field observation of yoga students and use factor analysis and item response theory to select the best items per dimension and to reduce the number of items in the measure. Phase IV will collect data on the new instrument and test the psychometric properties of the questionnaire (i.e., reliability and validity using data collected in Phases III and IV).

DETAILED DESCRIPTION:
The use of yoga for general health and wellness and for dealing with particular health conditions is increasing in the United States According to the National Health Interview Survey (NHIS) Alternative Medicine Supplement, the use of yoga increased significantly from 2002 to 2007 (NCCAM/Barnes, Bloom & Nahin, 2008), to 6.1% of the US population. In people dealing with health issues, the percent using yoga may be much higher (Birdee et al., 2008; NCCAM/Barnes et al., 2008). For example, in recent years, yoga has become a core complementary approach sought out by cancer patients and survivors of all cultural backgrounds in dramatically larger numbers (Mackenzie, Carlson, Munoz, & Speca, 2007).

Yoga interventions are being introduced for a variety of health conditions. Research evaluating these interventions remains inconclusive (NCCAM/Barnes et al., 2008) but preliminary results are promising. Many studies have reported evidence of superiority of yoga interventions relative to controls, although it is often difficult to determine the adequacy of the control condition. Reviewing the studies that compared yoga specifically to a physical exercise control condition, Ross and Thomas (2010) reported favorable findings for the impact of yoga on specific health conditions including cardiovascular disease (e.g., Raub, 2002), metabolic syndrome (e.g., Innes et al., 2005), diabetes (e.g., Upadhyay et al., 2008), cancer (see Bower et al., 2005) and anxiety (see Kirkwood et al., 2005). Similarly, a review of yoga interventions for chronic lifestyle-related diseases (Tekur et al., 2008) noted that yoga has been shown to be effective for treating osteoarthritis (Garfinkel et al., 1998), rheumatoid arthritis (Haslock et al., 1994), essential hypertension (Murugesan et al., 2000), bronchial asthma (Nagarathna et al., 1985; Vedanthan et al., 1998), irritable bowel syndrome (Taneja et al., 2004), diabetes (Singh et al., 2001), coronary artery disease (Manchanda et al., 2000), and depression (Woolery et al., 2004). Yoga has also been used in patients with chronic lower back pain (CLBP). Two randomized control trials on yoga for CLBP using Viniyoga (Sherman et al., 2005) and Iyengar yoga therapy (Williams et al., 2009) showed reduction in pain and functional disability relative to control groups. These studies contribute to the accumulating body of research evidence attesting to the positive health benefits of yoga. The recent NCCAM report indicates that, while promising, much more research evaluating these interventions is needed (NCCAM/Barnes et al., 2008). Currently, the content and substance of yoga remains a "black box" in that no studies have identified the effective ingredients of yoga. The proposed study will develop a tool to identify and quantify the components of yoga. The tool will thus allow researchers to link specific components of yoga to specific health outcomes such as pain, depression, functioning, etc.

ELIGIBILITY:
Inclusion Criteria:

* Yoga teachers, students, and researchers

Exclusion Criteria:

* Those who do not participate in regular (weekly) yoga practice

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Yoga teachers, students, and researchers.
Sampling Method: Non-Probability Sample
Enrollment: 1832 (Actual)
Dates: Start 2011-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
EPYQ Essential Properties of Yoga Questionnaire | Post yoga class in Phase IV
  The EPYQ is the survey that is being developed for this study to assess the essential properties of a yoga class or intervention

CONTACTS AND LOCATIONS:
Overall Officials: Erik Groessl, PhD, Principal Investigator — University of California, San Diego; Rani Elwy, PhD, Principal Investigator — Boston University; Susan Eisen, PhD, Principal Investigator — Boston University
Locations (1):
- Crystal Park, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No